CLINICAL TRIAL: NCT06114901
Title: Efficacy of Mobile-delivered Sleep Restriction Therapy for Treatment of Insomnia Disorder: Randomised Controlled Trial
Acronym: SleepFix
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X23-0371
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-10

CONDITIONS: Insomnia
Keywords: CBTi; Digital CBTi; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Online (digital), two-arm, open-label randomised clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research staff and Principal Chief Investigator will not be blinded to the study as they will be managing the online study directly which will lend itself to knowing which groups participants are allocated to. All other Investigators including data analysts will be blinded throughout the course of the trial and analysis of primary and secondary outcomes. Participants will not be blinded as they will know what treatment they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - SleepFix (Experimental): Participants will get access to a webpage and video which will show participants information about the dBTi SleepFix mobile application. This information will explain application download, usage concepts and frequently asked questions (FAQ). The intervention webpage will continue to be available for the participants throughout the intervention period for reference if necessary and be only accessible by this group. Participants will also be sent an email and/or text message with a direct link to iOS or Google play app stores to download the "SleepFix" mobile application. They will be provided a unique alphanumeric access code and instructed to enter this code to access the app program. Participants will be able to commence therapy immediately upon app onboarding.
  Interventions: Other: SleepFix
- Control - Sleep Health Education modules (Active Comparator): The participant will receive a link to three Sleep Health Education modules bi-weekly. All participants in the control group will gain access to the SleepFix mobile application upon completing their control period.
  Interventions: Other: Sleep health Education modules

INTERVENTIONS:
Other: SleepFix — SleepFix mobile application uses Sleep Retraining Therapy (SRT) which aims to reduce excess time spent in bed and reset sleep by matching time in bed (minimum of five and a half hours) to total sleep time (TST). There are four stages to the dBTi application and participants will progress based on completion of each stage. At the commencement of SleepFix application, participants enter sleep and bedtime data into the smartphone application for baseline referencing. These data are used to determine the sleep therapy based on a pre-determined algorithm that calculates optimum sleep efficiency.
  Arms: Intervention - SleepFix
Other: Sleep health Education modules — Three Sleep Health education modules that contain information about sleep hygiene and introduces strategies on how to reduce insomnia severity and increase sleep quality.
  Arms: Control - Sleep Health Education modules

SUMMARY:
The "SleepFix Study" is a clinical trial designed to evaluate the efficacy of mobile-delivered sleep restriction therapy (dBTi) in comparison to digital sleep health education (control) for treating insomnia disorder in adults aged 18 and above. The study is conducted entirely online, with 558 participants (279 in each group) and aims to determine the impact of the interventions on insomnia symptom severity, sleep metrics, subjective sleep quality, fatigue, anxiety, depressive symptoms, quality of life, medication usage, and workforce productivity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* Able to give informed online consent
* Insomnia Severity Index ≥ 12
* English fluency
* Access to a smartphone and willingness/proficiency to use a mobile application

Exclusion Criteria:

* Shift-workers (at least 2 night shifts a week between the hours of 8 pm to 8 am)
* Serious medical and/or psychiatric illnesses/disorders
* Previously diagnosed or suspected/high-risk of undiagnosed sleep disorders (e.g. REM Sleep Behaviour Disorder, Restless Leg Syndrome
* Currently receiving Cognitive Behavioural Therapy for insomnia (CBT-i)
* Operators of machinery that require high alertness (e.g. truck drivers, train drivers, pilots, etc)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-10-26 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia symptom severity change | 8 weeks
  Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 28) regarding symptoms over the past 2 weeks. Scores range from 0-28 with higher scores indicating greater insomnia symptom severity.

SECONDARY OUTCOMES:
Change in sleep-wake metrics | 8 weeks
  Sleep- wake metrics will be determined from the Pittsburgh Sleep Quality Index Score (PSQI) - a 19-item questionnaire with seven component scores derived from the responses, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0-21) where a score of 5 or more indicates poor sleep quality.
Daytime symptoms of fatigue | 8 weeks
  The Flinders Fatigue Scale (FFS) is a 7-item self-reported instrument designed to measure the level of subjective daytime fatigue experienced over the previous two weeks. 6-items consist of a 5-point Likert type scale ranging from "not at all" = 0 to "extremely" = 4. Item 5 uses a multiple-item checklist and is scored as a sum. All items are summed with total scores ranging from 0-31 with higher scores reflecting greater fatigue.
Change in anxiety scores | 8 weeks
  The General Anxiety Disorder-7 (GAD-7) is a 7-item self-administered scale used to assess the severity of generalised anxiety over the previous 2 weeks. It consists of a three-point Likert type scale for each item (ranging from "not at all" = 0 to "nearly every day" = 3). All items are summed with total scores ranging from 0-21 where 5, 10 and 15 indicate the cut-off scores for mild, moderate and severe anxiety, respectively.
Change in depressive symptom scores | 8 weeks
  The Patient Health Questionnaire-8 is an 8-item self-reported measure of depressive symptoms over the past 2 weeks. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
Change in quality of life scores | 8 weeks
  The EuroQol five-dimensional (EQ-5D) is a self-reported questionnaire which assesses 5 dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression and overall health. The 5 dimensions range from "1 = indicating no problem" - "5 = indicating unable to/extreme problems" and the overall score from 0 (worst health state imaginable) to 100 (best health state imaginable).
Treatment usability | 8 weeks
  The System Usability Scale (SUS) questionnaire is a 10-item survey that examines four dimensions of usability: useful- ness, ease of use, ease of learning, and satisfaction. It is scored out of a 100; scores closer to 100 means excellent usability while scores closer to 0 means worse usability.
Workforce productivity | 8 Weeks
  Participants will be asked short yes/no questions regarding the use of sleep medication in the previous two weeks.
Sleep medication usage | 8 weeks
  Participants will be asked short yes/no questions regarding taking sick leaves in the previous two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gordon, PhD, Principal Investigator — Macquarie University, Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No